CLINICAL TRIAL: NCT00121407
Title: A Randomized, Placebo-Controlled, Double-Masked, Multicenter, Phase III Study of the Effect of Visudyne Therapy in Occult With No Classic Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD): Visudyne in Occult (VIO)
Brief Title: Visudyne® in Occult (VIO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPD OCR 013 (VIO)
Record Dates: First submitted 2005-07-12; First posted 2005-07-21 (Estimated); Last update posted 2005-07-21 (Estimated); Status verified 2005-07

CONDITIONS: Macular Degeneration
Keywords: Age Related Macular Degeneration (AMD); Photodynamic Therapy (PDT); Visudyne
MeSH Terms: conditions — Macular Degeneration | interventions — Verteporfin; Injections

INTERVENTIONS:
Drug: Visudyne for injection

SUMMARY:
The purpose of this study is to demonstrate that Visudyne therapy in patients who have occult with no classic subfoveal choroidal neovascularization (CNV) lesions will, with an acceptable safety profile, significantly reduce the risk of vision loss compared with placebo (sham treatment).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double masked, multicenter, Phase III study. Patients will be stratified by study center and randomized to Visudyne therapy or placebo in a 2:1 ratio, respectively. Patients will receive either a single intravenous dose of Visudyne or placebo followed 15 minutes after the start of the infusion by light application. Follow-up visits will occur every three months (+/- 2 weeks) for the duration of the study. Re-treatment may be administered every three months (through the Month 21 visit) if evidence of CNV leakage is detected by fluorescein angiography (as judged by the Investigator).

At baseline and at each follow-up visit, patients will undergo the following assessments: ophthalmic examination, best-corrected visual acuity, color fundus photography, and fluorescein angiography. Indocyanine green (ICG) angiography will be conducted at baseline, Month 12, and Month 24. Optical coherence tomography (OCT) will be done at baseline, Month 3, Month 6, Month 12, and Month 24. Adverse events and concomitant medications will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients are men or women age 50 years or older.
* Patients must have occult CNV secondary only to AMD in the study eye, without any other concurrent retinal disease present that may also be associated with CNV (e.g., pathologic myopia, ocular histoplasmosis syndrome, etc.). In the case that both eyes are eligible, only one eye will be treated and the decision of which eye will be treated will be made between the patient and physician.
* Patients must have blood associated with the lesion or must have shown a progression of the disease within the preceding 3 months before randomization to treatment. For the purpose of this study, disease progression is defined as either:

  * a documented loss of vision (six or more letters with the ETDRS chart or at least three lines with a Snellen chart) using best-corrected visual acuity assessments; or
  * documented fluorescein angiographic evidence of a 10% increase in the lesion's greatest linear dimension.
* Patients must have lesions in the study eye with the following characteristics as determined by fluorescein angiography:

  * Evidence that occult CNV involves the geometric center of the foveal avascular zone;
  * The lesion has only occult CNV with no classic CNV;
  * The area of occult CNV must occupy at least 50% of the total lesion.
* Patients must have a best-corrected visual acuity score in the study eye between 73 and 34 letters (approximate Snellen equivalent of 20/40 to 20/200), inclusive. Visual acuity will be measured with an ETDRS chart using the procedure developed for the TAP/VIP studies.
* Patients must meet at least one of the following criteria:

  * CNV lesion ≤4 MPS disc areas;
  * Visual acuity score <65 letters.
* Female patients of child-bearing potential must not be pregnant or lactating, must have a negative pregnancy test (serum or urine) at baseline and must be practicing an adequate method of birth control. Acceptable methods of birth control include intrauterine device (IUD); oral, implanted or injected contraceptives; and barrier methods with spermicide.
* Patients must sign an approved informed consent that complies with relevant regulatory requirements prior to undergoing any study-related procedures.

Exclusion Criteria:

* Patients with a greatest linear dimension (GLD) of the entire lesion that exceeds 5400 microns
* Patients with a lesion size >6 MPS disc area (15.24 mm2)
* Patients with a CNV lesion size that is >4 MPS disc areas associated with a best-corrected visual acuity score that is >=65 letters (approximate Snellen equivalent of 20/50 or better) at the initial visit.
* Patients who have a known hypersensitivity/allergy to Visudyne, porfimer sodium, or other porphyrins; porphyria or other porphyrin sensitivity; or hypersensitivity to sunlight or bright artificial light.
* Patients who have the following in the study eye: a tear (rip) of the RPE; a vitelliform-like lesion of the outer retina (e.g., as in pattern dystrophies or basal laminar drusen); idiopathic parafoveal telangiectasis, retinal lesion anastomosis, or central serous retinopathy.
* Patients with a known allergy to fluorescein dye.
* Patients who have any additional ocular diseases which have irreversibly compromised or, during follow-up, could likely compromise the visual acuity of the study eye including amblyopia, elevated intraocular pressure (≥30 mm Hg), anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non proliferative diabetic retinopathy, proliferative diabetic retinopathy or cataract (lens or capsule) obscuring easy identification of the CNV lesion on biomicroscopy or fluorescein angiography.
* Patients who are unable to be photographed to document CNV, e.g., due to media opacity, cataract obscuring the CNV, allergy to fluorescein dye, or lack of venous access.
* Patients who have had treatment for CNV in the study eye with photodynamic therapy (PDT), transpupillary thermotherapy (TTT), or other local treatment (such as submacular surgery). Previous laser photocoagulation therapy is acceptable, provided it was not subfoveal.
* Patients who are participating in any other clinical study or are receiving, or have received any experimental systemic treatment for AMD (e.g., retinoic acid, thalidomide) or any other investigational new drug within 12 weeks prior to the start of study treatment.
* Patients who have undergone intraocular surgery within the last two months or Nd:YAG capsulotomy within the last month in the study eye.
* Patients who have a history of moderate to severe hepatic impairment (patients with this history may be included if laboratory tests are performed and results indicate that they are within the normal limits).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364
Dates: Start 2002-03; Study Completion 2005-08

PRIMARY OUTCOMES:
The primary efficacy variable is the patient responder rate. The patient responder rate has two definitions as described below:
• The proportion of patients who lose less than 15 letters (<3 lines) of best-corrected visual acuity in the study eye from baseline
• The proportion of patients who lose fewer than 30 letters (<6 lines) of best-corrected visual acuity in the study eye from baseline

SECONDARY OUTCOMES:
• The proportion of patients whose best-corrected visual acuity decreased to fewer than 34 letters (approximate Snellen equivalent of 20/200)
• Change from baseline in visual acuity score
• Cumulative proportion of patients who develop predominantly classic CNV in the study eye (identified by the Investigator and confirmed by a central reading center).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, MD, Study Director — QLT Inc.

REFERENCES:
- [Derived] Kaiser PK; Visudyne In Occult CNV (VIO) study group. Verteporfin PDT for subfoveal occult CNV in AMD: two-year results of a randomized trial. Curr Med Res Opin. 2009 Aug;25(8):1853-60. doi: 10.1185/03007990903038616. PMID 19530976
- See also: QLT website — http://www.qltinc.com